CLINICAL TRIAL: NCT06312371
Title: Intermittent Oro-esophageal Tube on Feeding Hesitancy in Stroke Patients: A Randomized Controlled Study
Brief Title: Intermittent Oro-esophageal Tube on Feeding Hesitancy in Stroke Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad (Other)
Responsible Party: Sponsor-Investigator, Muhammad, Research Director, Ahmadu Bello University Teaching Hospital
Organization: Ahmadu Bello University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Feeding Hesitancy
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Oro-esophageal Tube Feeding (Experimental): The group was given enteral nutritional support with Intermittent Oro-esophageal Tube according to the following procedure. The feeding content was formulated by the nutritionists based on the condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups
  Interventions: Device: Intermittent Oro-esophageal Tube Feeding
- Nasogastric Tube Feeding (Active Comparator): the group was given enteral nutritional support with Nasogastric Tube according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements.
  Interventions: Device: Nasogastric Tube Feeding

INTERVENTIONS:
Device: Intermittent Oro-esophageal Tube Feeding — Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm.
  Arms: Intermittent Oro-esophageal Tube Feeding
Device: Nasogastric Tube Feeding — Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the patient's cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time.
  Arms: Nasogastric Tube Feeding

SUMMARY:
The aim of this clinical trial is to compare Feeding Hesitancy of ischemic stroke patients who receive enteral nutrition support through either Intermittent Oro-esophageal Tube or Nasogastric Tube. Patients will be randomly assigned to either an observation group or a control group, with both groups receiving routine rehabilitation treatment. The observation group will receive enteral nutrition support through Intermittent Oro-esophageal Tube, while the control group will receive it through Nasogastric Tube. Researchers will then compare Feeding Hesitancy of the two groups.

DETAILED DESCRIPTION:
The study will last 15 days for each participant. The aim of this clinical trial is to compare Feeding Hesitancy of ischemic stroke patients who receive enteral nutrition support through either Intermittent Oro-esophageal Tube or Nasogastric Tube. Patients will be randomly assigned to either an observation group or a control group, with both groups receiving routine rehabilitation treatment. The observation group will receive enteral nutrition support through Intermittent Oro-esophageal Tube, while the control group will receive it through Nasogastric Tube. Researchers will then compare Feeding Hesitancy of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years;
* meeting the diagnostic criteria of stroke;
* any degree of dysphagia at admission;
* steady vital signs.

Exclusion Criteria:

* complicated with other neurological diseases;
* tracheostomy tube plugged;
* unfeasible to the support of parenteral nutrition;
* simultaneously suffering from liver, kidney failure, tumors, or hematological diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Swallowing Quality of Life questionnaire | day 1 and day 15
  Swallowing Quality of Life questionnaire was used to evaluate the quality of life, which consists of 44 items and divided into 11 main domains, including: overall satisfaction, understanding, diet, hydration, communication, respiratory issues, postoperative recovery, social impact, mental health, saliva control, and appearance. The maximum rough score was 220 points, which was converted into a standard percentage system in our study. As the scores increased, the quality of life was better.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Study Director — Site Coordinator of United Medical Group